CLINICAL TRIAL: NCT07059845
Title: A Phase 2, Open-Label, Randomized, Master Protocol Dose Optimization Study to Evaluate Safety and Efficacy of Multiple Treatment Combinations With Mirvetuximab Soravtansine in Subjects With Ovarian Cancer
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Multiple Treatment Combinations With Intravenous Mirvetuximab Soravtansine in Adult Participants With Ovarian Cancer
Acronym: FLORENZA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-709; 2025-521606-18 (Other: EU CT)
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Mirvetuximab Soravtansine; Bevacizumab; Carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — mirvetuximab soravtansine; Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Substudy 1 Arm A: Mirvetuximab Soravtansine (MIRV) Dose A (Experimental): Participants will receive dose A of MIRV with bevacizumab (Bev), as part of the approximately 40 month study duration.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Bevacizumab
- Substudy 1 Arm B: MIRV Dose B (Experimental): Participants will receive dose B of MIRV with Bev, as part of the approximately 40 month study duration.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Bevacizumab
- Substudy 1 Arm C: Bev (Experimental): Participants will receive Bev, as part of the approximately 40 month study duration.
  Interventions: Drug: Bevacizumab
- Substudy 2 Arm D: MIRV Dose A (Experimental): Participants will receive dose A of MIRV with carboplatin, followed by MIRV alone, as part of the approximately 31 month study duration.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Carboplatin
- Substudy 2 Arm E: MIRV Dose B (Experimental): Participants will receive dose B of MIRV with carboplatin, followed by MIRV alone, as part of the approximately 31 month study duration.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Carboplatin

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — Intravenous (IV) infusion
  Arms: Substudy 1 Arm A: Mirvetuximab Soravtansine (MIRV) Dose A; Substudy 1 Arm B: MIRV Dose B; Substudy 2 Arm D: MIRV Dose A; Substudy 2 Arm E: MIRV Dose B
Drug: Bevacizumab — IV Infusion
  Arms: Substudy 1 Arm A: Mirvetuximab Soravtansine (MIRV) Dose A; Substudy 1 Arm B: MIRV Dose B; Substudy 1 Arm C: Bev
Drug: Carboplatin — IV Infusion
  Arms: Substudy 2 Arm D: MIRV Dose A; Substudy 2 Arm E: MIRV Dose B

SUMMARY:
Ovarian cancer is a lethal disease with an estimated 310,000 new cases and 200,000 deaths experienced worldwide in 2020. The purpose of this study is to assess the adverse events and change in disease activity of mirvetuximab soravtansine with carboplatin, or bevacizumab (Bev), or bev alone in participants with ovarian cancer (OC). Participants must have confirmation of folate receptor alpha (FRa) positivity by the Ventana folate receptor 1 (FOLR1) Assay.

Mirvetuximab Soravtansine (MIRV) is an investigational drug for the treatment of OC. Participants will be assigned to 1 of 2 substudies and further into groups called treatment arms. In substudy 1, arms A-C, participants will receive 1 of 2 doses of MIRV with Bev, or Bev alone. In substudy 2, arms D and E, participants will receive 1 of 2 doses of MIRV with carboplatin, followed by MIRV alone. Approximately 320 participants will be enrolled in the study at 100 sites around the world.

Participants will receive intravenously (IV) infused MIRV with IV infused carboplatin, or IV infused Bev, or IV infused Bev alone. The total study duration will be approximately 40 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Substudy 1 and 2: Confirmed high or medium folate receptor alpha (FRa) expression by Ventana folate receptor 1 (FOLR1) Assay.
* Substudy 1 and 2: Participants must have an Eastern Cooperative Oncology Group performance status of 0 or 1.
* Substudy 1: Participants must have a confirmed diagnosis of Federation of Gynecology and Obstetrics (FIGO) Stage III or IV high-grade serous ovarian, primary peritoneal, or fallopian tube cancer.
* Substudy 1: Tumor must be confirmed HRD test negative (HRP), determined by a local homologous recombination deficient (HRD) test.
* Substudy 2: Participants must have a confirmed diagnosis of high-grade serous ovarian, primary peritoneal, or fallopian tube cancer.
* Substudy 2: Participants must have relapsed after 1 or 2 prior lines of platinum-based chemotherapy.
* Substudy 2: Participants must have platinum-sensitive disease defined as radiographic progression greater than 6 months from the last dose of platinum-based chemotherapy.
* Substudy 2: Participants must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (assessed by the investigator) at baseline.

Exclusion Criteria:

* Substudy 1: Participants with progressive disease (PD) while on triplet therapy or after the first day of their last triplet therapy cycle and before randomization.
* Substudy 1: Participants who receive an intervening dose of bevacizumab after the first day of their last triplet therapy cycle and before randomization.
* Substudy 1: Participants who received prior treatment with mirvetuximab soravtansine, any FRα-targeting agent, or any investigational agent.
* Substudy 2: More than 2 prior lines of chemotherapy. Lines of prior anticancer therapy are counted with the following considerations:
* Neoadjuvant +/- adjuvant therapies are considered 1 line of therapy if the neoadjuvant and adjuvant correspond to 1 fully predefined regimen; otherwise, they are counted as 2 prior regimens.
* Maintenance therapy (e.g., bevacizumab, PARP inhibitor) will be considered part of the preceding line of therapy (i.e., not counted independently).
* If a chemotherapeutic agent in a regimen is substituted with another during a course of treatment due to toxicity, it will be considered part of the proceeding line of therapy
* Prior hormonal therapy will not be counted as a separate line of chemotherapy (it will be counted as part of the prior systemic therapy regimen)
* Substudy 2: Participants who received prior treatment with mirvetuximab soravtansine or other FRα-targeting agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Substudy 1 and 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) (any grade, Grade >= 3) | Up to Approximately 40 Months
  TEAEs defined as any adverse event (AE) with the onset after the first dose of study drug until 30 days after the last dose of the study drug.
Substudy 1 and 2: Number of Participants with TEAEs Leading to Discontinuation | Up to Approximately 40 Months
  TEAEs defined as any adverse event (AE) with the onset after the first dose of study drug until 30 days after the last dose of the study drug.
Substudy 1 and 2: Number of Participants with Ocular Adverse Events (AEs) (any grade, Grade >= 2) | Up to Approximately 40 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Substudy 1 and 2: Overall Response (OR) as Assessed by the Investigator per RECIST v1.1 | Up to Approximately 40 Months
  OR is defined as achieving a best overall response of confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Substudy 1: Progression free survival (PFS) as Assessed by the Investigator per RECIST v1.1 | Up to Approximately 40 Months
  PFS is defined as the time from the date of randomization to the first occurrence of radiographic progression based on RECIST version 1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Substudy 1 and 2: CA-125 Response per Gynecologic Cancer Intergroup (GCIG) Criteria | Up to Approximately 40 Months
  CA-125 response per GCIG Criteria.
Substudy 1 and 2: Duration of Response (DOR) as Assessed by the Investigator per RECIST v1.1 | Up to Approximately 40 Months
  DoR is defined for confirmed responders as the time from the participants' initial response (CR or PR) to the first occurrence of radiographic progression per RECIST v1.1 or death from any cause.
Substudy 1 and 2: Number of Participants with Peripheral Neuropathy AEs (any grade, Grade ≥ 2) | Up to Approximately 40 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Substudy 1 and 2: Number of Participants with Pneumonitis/ Interstitial Lung Disease (ILD) (any grade) | Up to Approximately 40 Months
  ILD is defined by ILD standardized MedDRA query (SMQ) (broad) per investigator and determined per adjudication.
Substudy 2: PFS as Assessed by the Investigator per RECIST v1.1 | Up to Approximately 40 Months
  PFS is defined as the time from the date of randomization to the first occurrence of radiographic progression based on RECIST version 1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- Australia (6):
  - St. George Private Hospital /ID# 276570, Kogarah, New South Wales
  - Icon Cancer Centre Wesley /ID# 277199, Auchenflower, Queensland
  - Burnside War Memorial Hospital /ID# 277602, Adelaide, South Australia
  - Icon Cancer Centre Hobart /ID# 277688, Hobart, Tasmania
  - Monash Health - Monash Medical Centre /ID# 276984, Clayton, Victoria
  - Austin Hospital /ID# 276534, Melbourne, Victoria
- South Korea (4):
  - Seoul National University Hospital /ID# 276182, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 276266, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 276261, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 276194, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-709